CLINICAL TRIAL: NCT00387179
Title: Circadian Integration of Photic and Non-photic Stimuli
Brief Title: Effectiveness of Combining Light and Non-Light Treatments for Jet Lag and Sleep Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Kenneth P. Wright Jr., Ph.D., Associate Professor, University of Colorado
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 406; M01RR000051 (NIH); R01HL081761 (NIH)
Record Dates: First submitted 2006-10-11; First posted 2006-10-12 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Sleep Disorders, Circadian Rhythm
Keywords: Circadian Rhythm Sleep Disorders
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm | interventions — Melatonin; methylxanthine; Phototherapy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Dim Light Melatonin and/or methylxanthine (Experimental): Dim Light Melatonin and/or methylxanthine
  Interventions: Drug: Melatonin; Drug: Methylxanthine
- Placebo and Dim Light or bright light (Experimental): Placebo and Dim Light or bright light
  Interventions: Procedure: Light Therapy
- Bright light melatonin and/or methylxanthine (Experimental): Bright light, melatonin, and/or methylxanthine
  Interventions: Drug: Melatonin; Drug: Methylxanthine; Procedure: Light Therapy

INTERVENTIONS:
Drug: Melatonin — 5mg, pill, once
  Other Names: Life Extension Melatonin 5 mg
  Arms: Bright light melatonin and/or methylxanthine; Dim Light Melatonin and/or methylxanthine
Drug: Methylxanthine — 2.9 mg/kg, pill, once
  Arms: Bright light melatonin and/or methylxanthine; Dim Light Melatonin and/or methylxanthine
Procedure: Light Therapy — Bright light exposure
  Arms: Bright light melatonin and/or methylxanthine; Placebo and Dim Light or bright light

SUMMARY:
Jet lag and some sleep disorders are caused by a disruption in an individual's "internal clock." Understanding the most effective way to quickly re-adjust the body's internal clock will be beneficial for treating individuals with these conditions. This study will evaluate the combined effectiveness of light and non-light therapies at regulating sleep cycles and improving sleep quality.

DETAILED DESCRIPTION:
Circadian rhythm disorders are disruptions in an individual's circadian rhythm, or "internal body clock." This internal clock regulates the 24-hour cycle of biological processes in the body, including sleep and hormone production. Jet lag, delayed sleep phase syndrome, in which individuals fall asleep and wake up later than desired, and advanced sleep phase syndrome, in which individuals fall asleep and wake up earlier than desired, are all examples of circadian rhythm disorders. Because of the disruptive nature of these conditions, it is important to identify the quickest and most effective method for regulating the body and reestablishing normal sleep patterns. Light therapy, in which individuals are exposed to bright, artificial light, is currently used to treat these disorders. Melatonin, a hormone that regulates circadian rhythms, and methylxanthines, a class of stimulant medications, are other common non-light treatments. While each of these individual treatments has been proven effective, little is known about the combined effect of light and non-light treatments. The purpose of this study is to evaluate the safety and effectiveness of light therapy, melatonin, and methylxanthine, alone and in combination, at regulating circadian rhythms and improving sleep quality and cognitive function.

This study will enroll healthy individuals. Participants will first attend two screening visits, which will include a review of medical, psychiatric, and sleep histories; vital sign measurements; blood and urine collection; a physical examination; and an electrocardiogram. For 1 week, participants will record sleep habits in a diary and by telephone. They will also wear a device that monitors activity and light exposure levels. Eligible participants will then attend four 5-day inpatient visits at the Sleep and Chronobiology Laboratory at the University of Colorado at Boulder. During each of the four visits, participants will be randomly assigned to one of the following four treatments:

* Dim light therapy and placebo
* Bright light therapy and placebo
* Dim light therapy, melatonin, and methylxanthines
* Bright light therapy, melatonin, and methylxanthines

At each visit, participants will receive a different treatment. During these visits, participants will remain awake for up to 40 hours at a time, while their eye movements, and brain, muscle, heart, and breathing activity are monitored. Urine and saliva will be collected, and participants will undergo various cognitive performance testing measures. At 3-week intervals between each visit, participants will record sleep habits and will wear the activity and light exposure monitoring device. A sleep diary will also be maintained by participants for 3 weeks following the end of the last visit.

ELIGIBILITY:
Inclusion Criteria:

* In good general health, as determined by blood chemistries, urine toxicology, physical examination, and medical and psychiatric history

Exclusion Criteria:

* History of any current or chronic disease, including any of the following:

  1. Chronobiologic disorders
  2. Sleep disorders
  3. Cardiovascular disorders
  4. Respiratory disorders
  5. Kidney and urinary tract disorders
  6. Infectious diseases
  7. Gastrointestinal disorders
  8. Immune system disorders
  9. Connective tissue and joint disorders
  10. Hematopoietic disorders
  11. Neoplastic diseases
  12. Endocrine and metabolic diseases
  13. Neurologic disorders
* Current or past history of drug abuse
* Pregnant or breastfeeding
* Current oral contraceptive use

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2006-10; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Circadian phase, as measured by the shift of the endogenous melatonin rhythm (measured during each inpatient visit) | 24 hour

SECONDARY OUTCOMES:
Circadian phase, as measured by the shift of the endogenous temperature rhythm | 24 hour
Sleep quality, as measured by wakefulness after sleep onset (electroencephalogram [EEG] defined wakefulness after 10 minutes of consecutive sleep) and number of awakenings | overnight
Cognitive function, as measured by daytime sleepiness, reaction time, and mood and well being (all measured during each inpatient visit) | 24 h and daytime

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth P. Wright, PhD, Principal Investigator — University of Colorado at Boulder
Locations (1):
- Sleep and Chronobiology Laboratory, Boulder, Colorado, United States

REFERENCES:
- [Background] Duffy JF, Wright KP Jr. Entrainment of the human circadian system by light. J Biol Rhythms. 2005 Aug;20(4):326-38. doi: 10.1177/0748730405277983. PMID 16077152
- [Background] Wright KP Jr, Gronfier C, Duffy JF, Czeisler CA. Intrinsic period and light intensity determine the phase relationship between melatonin and sleep in humans. J Biol Rhythms. 2005 Apr;20(2):168-77. doi: 10.1177/0748730404274265. PMID 15834113
- [Background] Gronfier C, Wright KP Jr, Kronauer RE, Jewett ME, Czeisler CA. Efficacy of a single sequence of intermittent bright light pulses for delaying circadian phase in humans. Am J Physiol Endocrinol Metab. 2004 Jul;287(1):E174-81. doi: 10.1152/ajpendo.00385.2003. Epub 2004 Mar 23. PMID 15039146
- [Background] Barger LK, Wright KP Jr, Hughes RJ, Czeisler CA. Daily exercise facilitates phase delays of circadian melatonin rhythm in very dim light. Am J Physiol Regul Integr Comp Physiol. 2004 Jun;286(6):R1077-84. doi: 10.1152/ajpregu.00397.2003. Epub 2004 Mar 18. PMID 15031136
- [Background] Wright KP Jr, Czeisler CA. Absence of circadian phase resetting in response to bright light behind the knees. Science. 2002 Jul 26;297(5581):571. doi: 10.1126/science.1071697. No abstract available. PMID 12142528
- [Background] Wright KP Jr, Hughes RJ, Kronauer RE, Dijk DJ, Czeisler CA. Intrinsic near-24-h pacemaker period determines limits of circadian entrainment to a weak synchronizer in humans. Proc Natl Acad Sci U S A. 2001 Nov 20;98(24):14027-32. doi: 10.1073/pnas.201530198. PMID 11717461
- [Background] Wright KP Jr, Myers BL, Plenzler SC, Drake CL, Badia P. Acute effects of bright light and caffeine on nighttime melatonin and temperature levels in women taking and not taking oral contraceptives. Brain Res. 2000 Aug 11;873(2):310-7. doi: 10.1016/s0006-8993(00)02557-9. PMID 10930561
- [Background] Wright KP Jr, Badia P, Myers BL, Plenzler SC, Hakel M. Caffeine and light effects on nighttime melatonin and temperature levels in sleep-deprived humans. Brain Res. 1997 Jan 30;747(1):78-84. doi: 10.1016/s0006-8993(96)01268-1. PMID 9042530
- See also: Click here for the University of Colorado at Boulder Sleep and Chronobiology Laboratory web site — http://www.colorado.edu/intphys/research/sleep.html